CLINICAL TRIAL: NCT01337297
Title: Treatment of Crack-cocaine Addiction Through Cognitive Neuromodulation of the Prefrontal Cortex Produced by Transcranial Direct Current Stimulation.
Brief Title: Prefrontal Cortex Stimulation as Treatment for Crack-cocaine Addiction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Harvard University (Other); University of Göttingen (Other)
Responsible Party: Principal Investigator, Ester Miyuki Nakamura-Palacios, MD, PhD, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP-UFES 296/10
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Cocaine Addiction; Cocaine-related Disorder; Executive Dysfunction
Keywords: crack cocaine; addiction; tDCS; ERP; P300; attention; inhibitory control; working memory
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Transcranial Direct Current Stimulation; Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham-tDCS (Placebo Comparator): the electrodes are positioned in the same manner as the active-tDCS, activated for 20 s (time to climb ramp of the current until reach the current intensity used in the experiment), enough to produce the sensation of itch, and turned off until the end of the session.
  Interventions: Device: transcranial Direct Current Stimulation
- active-tDCS (Experimental): low-intensity transcranial Direct Current Stimulation (tDCS)applied over the dorsolateral prefrontal cortex
  Interventions: Device: transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial Direct Current Stimulation — transcranial Direct Current Stimulation (tDCS) will be applied by electrodes (5 x 7 cm2), with intensity of 2 mA, during 20 min, with cathode over the left dorsolateral prefrontal cortex (F3 site) and anode placed in the contralateral dorsolateral prefrontal cortex (F4 site).
  Other Names: brain stimulation; non-invasive brain stimulation

SUMMARY:
The use of crack-cocaine is growing at alarming rate in our country and it is absolutely worrisome the fast establishment of addiction to it. Its immediate effects, that are intense and extremely fleeting, increase dramatically the probability of this drug to be consumed again, settling quickly down the loss of control and the compulsive use, turning the effects of this drug highly addictive. Parallel to this process, brain damages are quickly established, progressing to severe impairments of frontal functions, leading to the lack of cognitive control that feeds back and aggravates the dependence, and hampers any therapeutic approach. The existing treatments have not proved to be satisfactory yet. Thus, considering that a new modality of treatment, based on the neuromodulation induced by noninvasive brain stimulation, has been useful in treating various neuropsychiatric conditions, this study will examine the potential beneficial effects of repeated transcranial Direct Current Stimulation over the left dorsolateral prefrontal cortex in the treatment of crack-cocaine addiction.

DETAILED DESCRIPTION:
Forty subjects between 18 and 60 years old, both genders, with a diagnosis of dependence on crack-cocaine, evaluated for the first time at the Center for Psychosocial Care for Alcohol and Other Drugs (CAPS-AD, in Portuguese) in the municipality of Serra, ES, Brazil, will be invited to participate in this study. After triage, following the inclusion and exclusion criteria, they will be informed in details about the experimental protocol and, if they agree to participate, it will be required to sign an Informed Consent. It Will be applied a structured anamnesis, made a psychiatric clinical and physical examination. The treatment will be started with regular medications for abstinence and comorbidities and psychosocial approaches usually done in the CAPS-AD. After selected they will be referred to the Laboratory of Cognitive Science and Neuropsychopharmacology of the Postgraduate Program in Physiological Sciences from Health Sciences Center of Federal University of Espírito Santo where they will be semi-randomly (matched for age, gender and sociodemographic characteristics) distributed into two different groups: (A) sham-tDCS (n = 20) and (B) active-tDCS (n = 20); and they will follow for 10 applications in daily sessions, excepting on weekends, of transcranial direct current stimulation (tDCS, 5 x 7 cm2, 2 mA, 20 min) over the left dorsolateral prefrontal cortex or sham procedure. Event-related potentials (ERP) will be recorded before, during and after brain stimulation or sham procedure under random presentation of three related images and three non-related images to crack use. The compulsive behavior will be evaluated before and after the ERP records. Cognitive tests which assess mental function, frontal function, visuospatial and verbal working memory, inhibition, and conflict resolution will be performed. The depression will be assessed during the treatment, and the addicted subjects will be evaluated once a week for four consecutive weeks after a series of applications of sham-tDCS or active-tDCS.

ELIGIBILITY:
Inclusion Criteria:

* fulfill the criteria for the crack-dependence syndrome, based on criteria of the International Classification of Diseases on its 10th version;
* all users and addicts who make use of crack-cocaine alone or in combination with other drugs (alcohol, nicotine, caffeine, cannabis, etc.), or who have psychiatric comorbidities (anxiety, depression, etc.)
* must be clinically stable and not requiring hospitalization;
* should be clinically suitable for the treatment proposed in this study;
* need to be able to read, write and speak Portuguese

Exclusion Criteria:

* should not present current or past illnesses that may be aggravated during treatment;
* may not show abnormalities in laboratory tests which suggest a deterioration of its physical condition for participation in the study;
* individuals who have some metal in the brain or skull (chips, fragments, pins, etc. - except titanium);
* history of epilepsy, severe brain trauma, cochlear implant, cardiac pacemaker or intracardiac metal apparatus);
* pregnants.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ester M Nakamura-Palacios, MD, PhD, Principal Investigator — Federal University of Espírito Santo
Locations (1):
- Laboratory of Cognitive Sciences and Neuropsychopharmacology, Post-Graduation Program in Physiologycal Sciences, Health Sciences Center, Federal University of Espírito Santo, Vitória, Espírito Santo, Brazil

REFERENCES:
- [Background] Aharonovich E, Nunes E, Hasin D. Cognitive impairment, retention and abstinence among cocaine abusers in cognitive-behavioral treatment. Drug Alcohol Depend. 2003 Aug 20;71(2):207-11. doi: 10.1016/s0376-8716(03)00092-9. PMID 12927659
- [Background] Aharonovich E, Hasin DS, Brooks AC, Liu X, Bisaga A, Nunes EV. Cognitive deficits predict low treatment retention in cocaine dependent patients. Drug Alcohol Depend. 2006 Feb 28;81(3):313-22. doi: 10.1016/j.drugalcdep.2005.08.003. Epub 2005 Sep 19. PMID 16171953
- [Background] Boggio PS, Sultani N, Fecteau S, Merabet L, Mecca T, Pascual-Leone A, Basaglia A, Fregni F. Prefrontal cortex modulation using transcranial DC stimulation reduces alcohol craving: a double-blind, sham-controlled study. Drug Alcohol Depend. 2008 Jan 1;92(1-3):55-60. doi: 10.1016/j.drugalcdep.2007.06.011. Epub 2007 Jul 19. PMID 17640830
- [Background] Boggio PS, Rigonatti SP, Ribeiro RB, Myczkowski ML, Nitsche MA, Pascual-Leone A, Fregni F. A randomized, double-blind clinical trial on the efficacy of cortical direct current stimulation for the treatment of major depression. Int J Neuropsychopharmacol. 2008 Mar;11(2):249-54. doi: 10.1017/S1461145707007833. Epub 2007 Jun 11. PMID 17559710
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Franco GM. [The cognitive potential in normal adults]. Arq Neuropsiquiatr. 2001 Jun;59(2-A):198-200. Portuguese. PMID 11400024
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Derived] Conti CL, Nakamura-Palacios EM. Bilateral transcranial direct current stimulation over dorsolateral prefrontal cortex changes the drug-cued reactivity in the anterior cingulate cortex of crack-cocaine addicts. Brain Stimul. 2014 Jan-Feb;7(1):130-2. doi: 10.1016/j.brs.2013.09.007. Epub 2013 Oct 12. PMID 24139147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We started to recruit patients in 2011 in drug dependence specialized public outpatient service.
Pre-assignment Details: Of 70 patients, 20 filling including criteria and without excluding criteria were recruited. The remaining 50 either refused to participate or accepted but never showed up to the researcher center.
Groups:
- Active-tDCS: low-intensity transcranial Direct Current Stimulation (tDCS)applied over the dorsolateral prefrontal cortex
  transcranial Direct Current Stimulation : transcranial Direct Current Stimulation (tDCS) will be applied by electrodes (5 x 7 cm2), with intensity of 2 mA, during 20 min, with cathode over the left dorsolateral prefrontal cortex (F3 site) and anode placed in the contralateral dorsolateral prefrontal cortex (F4 site).
- Sham-tDCS: the electrodes are positioned in the same manner as the active-tDCS, activated for 20 s (time to climb ramp of the current until reach the current intensity used in the experiment), enough to produce the sensation of itch, and turned off until the end of the session.
  transcranial Direct Current Stimulation : transcranial Direct Current Stimulation (tDCS) will be applied by electrodes (5 x 7 cm2), with intensity of 2 mA, during 20 min, with cathode over the left dorsolateral prefrontal cortex (F3 site) and anode placed in the contralateral dorsolateral prefrontal cortex (F4 site).
Period: Overall Study
Arm/Group | Active-tDCS | Sham-tDCS
Started | 11 | 9
Completed | 6 | 3
Not Completed | 5 | 6
Not completed — They entered to single anodal tDCS | 4 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active-tDCS | Sham-tDCS | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (7.3) | 28.3 (5.0) | 29.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Brazil | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Abstinence
Description: abstinence to the use of crack-cocaine up to 3 months after the completion of two-weeks of treatment sessions with active-tDCS or sham-tDCS.
Time Frame: Two days after the end of tDCS treatment (one session every other day, 5 sessions), that is, on the 12nd day from the beginning.
Measure: Number; unit: percentage of participants
Arm/Group | Active-tDCS | Sham-tDCS
Number analyzed (Participants) | 7 | 6
percentage of participants | 71.4 | 16.6

2. Secondary Outcome: Intensity of the Urge to the Use of Crack-cocaine
Description: The intensity of craving will be examined by a short scale, the Brief Cocaine Craving Questionnaire.
Time Frame: before and after ERP in two weekly sessions over two weeks
Reporting Status: Not Posted

3. Secondary Outcome: Event Related Potentials
Description: Event Related Potentials (ERPs) elicited by random presentation of three related images and three non-related images to crack use every Monday and Friday over the two-weeks period of active-tDCS or sham-tDCS.
Time Frame: twice a week over two consecutive weeks during the treatment
Reporting Status: Not Posted

4. Secondary Outcome: Cognitive Tests
Description: Cognitive tests are comprised by frontal assessment battery (FAB), Mini-Mental Status Examination (MMSE), verbal n-back task, visuospatial n-back task, go/no-go test.
Time Frame: Before the first experimental session, in the middle of the protocol and two days after the last experimental session
Reporting Status: Not Posted

5. Secondary Outcome: State of Depression
Description: It will be applied Hamilton Scale for Depression, a structured multiple choice questionnaire used to assess the severity of the symptoms of depression. It will be applied with cognitive tests.
Time Frame: Before the first experimental session, in the middle of the treatment and after the last experimental session.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Active-tDCS | Sham-tDCS
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Crack-cocaine is highly addictive, extremely difficult to treat and with high dropouts. 7 subjects started with anodal DLPFC tDCS showing high relapses (not shown). The remaining 13 subjects tested with bilateral DLPFC tDCS or sham were considered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No